CLINICAL TRIAL: NCT04060628
Title: Expanded Access to NanoDoce
Status: No longer available | Type: Expanded Access
Sponsor: NanOlogy, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: NANODOCE-EA
Record Dates: First submitted 2019-08-14; First posted 2019-08-19 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Urogenital Neoplasms
MeSH Terms: conditions — Urogenital Neoplasms | interventions — Powders; Suspensions; Docetaxel

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: NanoDoce (sterile nanoparticulate docetaxel) Powder for Suspension
  Other Names: docetaxel

SUMMARY:
NanOlogy may consider offering expanded access to NanoDoce for patients who do not meet the enrollment criteria of clinical trials in progress.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult